CLINICAL TRIAL: NCT01449032
Title: MesenchYmal STROMAL CELL Therapy in Patients With Chronic Myocardial Ischemia (MyStromalCell Trial)
Acronym: MyStromalCell
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, JKastrup, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MyStromalCell
Record Dates: First submitted 2011-10-06; First posted 2011-10-07 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Ischemic Heart Disease
Keywords: Patients
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSC (Active Comparator): Adipose derived stem cells
  Interventions: Biological: MSC
- Saline (Placebo Comparator)
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: MSC — No of cells after culture expansion
  Other Names: Adipose derived stem cells; Mesenchymal stromal cells; Mesenchymal stem cells
  Arms: MSC
Biological: Saline — 3 cc saline
  Arms: Saline

SUMMARY:
Coronary artery disease (CAD) is the most common cause of death and a major cause of hospital admissions for acute chest pain. In spite of improved treatments still many patients with CAD have daily attacks of severe chest pain and severely reduced life quality.

The investigators have established a double-blind placebo-controlled trial in patients with CAD to test efficacy and safety of treatment with adipose derived stem cells to improve perfusion in the heart muscle and exercise capacity, and reduce the patient's symptoms.

DETAILED DESCRIPTION:
In an open single centre pilot study we have evaluated the safety and efficacy of MSC treatment to improve heart muscle perfusion in patients with chronic CAD. Patients treated with MSCs had significant increased exercise capacity, reduction in angina, angina attacks and medication and in life quality at 6 months follow-up. For all the parameters there was a tendency towards improved outcome with increasing number of cells. The treatment with MSCs was safe.

The investigators have now established a double-blind placebo-controlled trial in patients with CAD to test efficacy and safety of treatment with MSCs to improve perfusion in the heart muscle and exercise capacity, and reduce the patient's symptoms.

ELIGIBILITY:
Inclusion Criteria:

* CCS III - IV
* Coronary artery stenosis/occlusion not treatable with invasive procedures
* LVEF > 40%
* ETT between 2 - 10 min

Exclusion Criteria:

* Valvular heart disease
* FEV1 < 1
* Severe systemic disease
* Acute coronary syndrome > 2 months

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Exercise test | 6 months

SECONDARY OUTCOMES:
Clinical evaluation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kastrup, MD Professor, Principal Investigator — Department of Cardiology, Rigshospitalet
Locations (1):
- Rigshospitalet University Hospital Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Qayyum AA, Mathiasen AB, Helqvist S, Jorgensen E, Haack-Sorensen M, Ekblond A, Kastrup J. Autologous adipose-derived stromal cell treatment for patients with refractory angina (MyStromalCell Trial): 3-years follow-up results. J Transl Med. 2019 Nov 12;17(1):360. doi: 10.1186/s12967-019-2110-1. PMID 31711513
- [Derived] Qayyum AA, Mathiasen AB, Mygind ND, Kuhl JT, Jorgensen E, Helqvist S, Elberg JJ, Kofoed KF, Vejlstrup NG, Fischer-Nielsen A, Haack-Sorensen M, Ekblond A, Kastrup J. Adipose-Derived Stromal Cells for Treatment of Patients with Chronic Ischemic Heart Disease (MyStromalCell Trial): A Randomized Placebo-Controlled Study. Stem Cells Int. 2017;2017:5237063. doi: 10.1155/2017/5237063. Epub 2017 Dec 3. PMID 29333165